CLINICAL TRIAL: NCT02495415
Title: Phase II Trial of Intravenous Fenretinide (N-(4-hydroxyphenyl) Retinamide, 4-HPR) Emulsion for Patients With Relapsed/Refractory Peripheral T-cell Lymphomas (PTCL)
Brief Title: Trial of Intravenous Fenretinide Emulsion for Patients With Relapsed/Refractory Peripheral T-cell Lymphomas
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CerRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEN T-14
Record Dates: First submitted 2015-07-07; First posted 2015-07-13 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Fenretinide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fenretinide emulsion (Experimental): Patients enrolled will receive 600 mg fenretinide/m2/day on Day 1, followed by 1200 mg fenretinide/m2/day on Days 2 - 5 as a continuous intravenous infusion via central line over 5 days. Cycles are repeated every 3 weeks.
  Interventions: Drug: Fenretinide

INTERVENTIONS:
Drug: Fenretinide — Fenretinide intravenous emulsion administered as a continuous intravenous infusion for 5 days, once every 3 weeks in relapsed/refractory PTCL patients.
  Other Names: 4-HPR; (N-(4-hydroxyphenyl) retinamide

SUMMARY:
This study addresses the hypothesis that intermittent treatment with fenretinide intravenous emulsion will induce objective responses in patients with relapsed or refractory Peripheral T-cell Lymphoma (PTCL) who have failed at least one prior systemic therapy and will result in acceptable toxicities.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single arm efficacy and safety study in patients with relapsed or refractory peripheral T-cell lymphoma, who have failed at least one prior system therapy.

Approximately 140 patients will be enrolled. Patients will be treated with fenretinide (4-HPR) intravenous emulsion administered as a continuous intravenous infusion for 5 days, once every 3 weeks until there is disease progression or unmanageable treatment-related toxicities.

The primary study endpoint is objective response rate (ORR). Responses will be categorized using criteria established by the International Harmonization Project on Lymphoma. Safety will be evaluated during the study and for 30 days after the last administration of study drug. Adverse events and laboratory studies will be graded according to NCI-CTCAE v. 4.03.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years with histologically or cytologically confirmed Peripheral T-cell lymphoma (PTCL)
* Diseases refractory/relapsed after one or more systemic cytotoxic therapies; patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
* Patients with an ECOG performance status of 0, 1, or 2, and estimated survival of > 12 weeks.
* Patients with at least ONE of the following sites of measurable disease according to International Workshop Criteria87: A) Measurable tumor on MRI or CT scan. Measurable is defined as at least one lesion 20 mm in at least one dimension; for spiral CT, measurable is defined as 10 mm in at least one dimension. For patients with persistent disease, a biopsy of bone marrow, or bone, or a soft tissue site, must have demonstrated viable tumor. If lesion was radiated, biopsy must have been done at least 4 weeks after radiation completed. B) Bone marrow with tumor cells seen on routine morphology (not by NSE staining only) of bilateral aspirate and/or biopsy on one bone marrow sample, except for patient who tested positive subsequent to their last treatment regimen or patients who had a negative marrow within three months of study entry.

Exclusion Criteria:

* Unable to give written informed consent
* Patients who have received chemotherapy within 3 weeks of first fenretinide treatment, or who have received investigational drugs within 6 weeks of first fenretinide treatment. Patients must have otherwise recovered from toxicities of prior therapy.
* Patient is not eligible if radiation was given to the only site of measurable disease unless there has been subsequent disease progression at that site, or a biopsy of that site showed viable tumor at least 4 weeks after radiation was completed. Patients must not have received small field (focal) radiation for a minimum of 2 weeks prior to study entry. A minimum of 6 weeks is required following prior large field radiation therapy (i.e. TBI, craniospinal therapy, whole abdomen, total lung, > 50% marrow space)
* Patients who have uncontrolled systemic infections, coagulation disorders, or other major medical illnesses of the cardiovascular or respiratory systems.
* Patients with any active hepatitis infections.
* Growth factor(s): Must not have received any hematopoetic growth factors within 7 days of study entry.
* Organ Transplant: Patients may NOT be the recipients of an organ transplant.
* Women who are pregnant and/or lactating.
* Patients who have had major non-biopsy surgery in the last 20 days.
* CNS lesions: A) Patients with CNS parenchymal or meningeal-based lesions that are present at study entry are NOT eligible due to concerns regarding toxicity attribution. B) Who have active CNS disease or a history of cranial irradiation are excluded due to concerns regarding toxicity attribution. Patients with previously treated leptomeningeal disease or brain metastases without evidence of remaining tumor by PET, MRI scan, or spinal fluid will be eligible; however such patients currently taking steroids as prophylaxis against seizures are not eligible.
* Patients with documented allergy to egg products.
* Known history of, or positive test result for human immunodeficiency virus (HIV) infection.
* Patients with fasting serum triglycerides > 300 and/or with hypertriglyceridemia requiring medication (but not patients with hypercholesterolemia: patients with hypercholesterolemia with or without medication are eligible).
* Patients concurrently taking the following drugs are excluded: antioxidants, herbal or other alternative therapy medications, vitamin supplements (especially vitamins A, C, and E) other than at standard multivitamin doses, cyclosporine A or analogue; verapamil; tamoxifen or analogue, ketoconazole, chlorpromazine; RU486; indomethacin; or sulfinpyrazone, tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, and amiodarone. If the patients discontinue usage of the above drugs, they can be eligible for enrollment into the study (screening visit) one week or 5-half lives of the drug in question, whichever is the longer, after the discontinuation. For patients requiring any of these medications, entry is permissible only with permission from the medical monitor.
* Patients with poorly controlled diabetes mellitus with fasting serum glucose concentration over 200 mg/dl or a hemoglobin A1C over 7.5%.
* Patients with any known significant cardiac abnormality.
* Patients with uncontrolled hypertension.
* Participation in any other investigational treatment within the 6 weeks prior to enrollment or concurrent with this study.
* Patients with an identified familial hyperlipidemia disorder.
* Patients with documented allergy to soy products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Objective tumor responses will be measured and recorded during the two weeks following the completion of the drug infusion of every even-numbered treatment cycle until the patient is removed from the study.

SECONDARY OUTCOMES:
Safety and tolerability profile will be assessed by adverse events which will be graded according to NCI-CTCAE v. 4.03. | monitored from start of initial therapy until 30 days after the patient is removed from study therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kerry M. Barnhart, Ph.D., Study Director — CerRx, Inc.
Locations (11):
- United States (11):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Bon Secours Saint Francis Cancer Center, Greenville, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas, Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mohrbacher AM, Yang AS, Groshen S, Kummar S, Gutierrez ME, Kang MH, Tsao-Wei D, Reynolds CP, Newman EM, Maurer BJ. Phase I Study of Fenretinide Delivered Intravenously in Patients with Relapsed or Refractory Hematologic Malignancies: A California Cancer Consortium Trial. Clin Cancer Res. 2017 Aug 15;23(16):4550-4555. doi: 10.1158/1078-0432.CCR-17-0234. Epub 2017 Apr 18. PMID 28420721